CLINICAL TRIAL: NCT04933084
Title: Evaluation of Pre-operative Education Modalities to Decrease Opioid Use in Prostate Cancer Patients: A Prospective Randomized Control Trial
Brief Title: Pre-operative Education Modalities to Decrease Opioid Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Una Lee, Staff Urologist, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRP20107
Record Dates: First submitted 2021-06-11; First posted 2021-06-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Prostatectomy; Opioid-Related Disorders
Keywords: Opioid Education; Post-operative Opioid Use
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Triple-armed randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): During their pre-operative visit, the usual care group will undergo usual pre-surgery patient education care dependent on their provider.
- Text Handout (Experimental): This group will receive limited opioid analgesia in conjunction with pre-operative education in the form of a text handout.
  Interventions: Behavioral: Pre-operative Opioid Education
- Text handout and Pre-recorded Video (Experimental): This group will receive limited opioid analgesia in conjunction with pre-operative education in the form of a text handout AND pre-recorded video.
  Interventions: Behavioral: Pre-operative Opioid Education

INTERVENTIONS:
Behavioral: Pre-operative Opioid Education — The pre-operative education in the text handout and pre-recorded video will include the topics of:
  1. Description of expected postoperative pain after robotic prostatectomy and typical opioid consumption after RARP.
  2. Efficacy of non-opioid multimodal analgesia and recommendation to take nonopioid alternatives prior to prescribed opioids.
  3. Adverse short- and long-term effects of opioids including nausea, vomiting, sedation, hypoventilation, hypotension, dizziness, constipation, depression, and addiction.
  Arms: Text Handout; Text handout and Pre-recorded Video

SUMMARY:
This is a triple-armed, randomized, controlled, non-blinded trial to study the effect of preoperative patient education in conjunction with a limited opioid peri-operative analgesia program on post-operative opioid use following radical prostatectomy. Patients will be randomized into three education arms: usual care (variable provider-dependent education), text handout, or text handout and pre-recorded video. The impact of patient education on outcomes of in-hospital, post-discharge, and persistent opioid use will be studied.

DETAILED DESCRIPTION:
This is a triple-armed, randomized, controlled, non-blinded trial that will be conducted at Virginia Mason Medical Center (VMMC). Men of age 18 or older undergoing robotic assisted radical prostatectomy (RARP) for prostate cancer will be approached to participate in the study. Recruited patients will be randomized into three main groups based upon opioid education given to the patient before surgery: usual care group, text handout group, and text handout with pre-recorded video group.

During their pre-operative visit, the usual care group will undergo usual pre-surgery patient education care dependent on their provider. The study group will receive additional standardized pre-operative education including the topics of:

1. Description of expected postoperative pain after robotic prostatectomy and typical opioid consumption after RARP.
2. Efficacy of non-opioid multimodal analgesia and recommendation to take nonopioid alternatives prior to prescribed opioids.
3. Adverse short- and long-term effects of opioids including nausea, vomiting, sedation, hypoventilation, hypotension, dizziness, constipation, depression, and addiction.

Patients in both usual care and study groups will receive standardized multimodal analgesia program with minimal opioids used.

Primary outcomes measured will include in-hospital and post-discharge opioid use, pain levels and time to return of bowel function. Secondary outcomes will include daily measures of patient satisfaction and quality of life, feeling of preparedness to manage post-operative pain, as well as incidence of prolonged opioid use at 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Undergoing RARP at VMMC
* Consent to participate in the study

Exclusion Criteria:

* Long-term opioid use defined as use of opioids on most days for >3 months
* History of drug or alcohol dependence
* Concurrent surgery during radical prostatectomy
* History of allergy to opioid analgesics, NSAIDs, acetaminophen or local anesthetics
* Inability or unwillingness to give written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
In-hospital opioid use | Immediately after the intervention/procedure/surgery
  Morphine equivalents used in the hospital will be calculated.
Post-discharge opioid use | Immediately after the intervention/procedure/surgery
  Patient-reported number of opioid pills used after discharge (daily questionnaire).
Post-operative pain | Immediately after the intervention/procedure/surgery
  Average pain over the course of today. (0=no pain, 5=moderate pain, 10=severe pain)
Return of bowel function | Immediately after the intervention/procedure/surgery
  Patient-reported return of bowel function as time in days to first flatus and first bowel movement.

SECONDARY OUTCOMES:
Satisfaction with undergoing the surgery | Immediately after the intervention/procedure/surgery
  Satisfaction with undergoing the surgery. (1=extremely dissatisfied, 10=extremely satisfied)
Quality of life after undergoing surgery | Immediately after the intervention/procedure/surgery
  Quality of life after the surgery. (1=worst possible QOL, 10=best possible QOL)
Prolonged post-operative opioid use | Up to 24 weeks
  Incidence of prolonged postoperative opioid use defined by the American Society of Interventional Pain Physicians Guidelines as continued use beyond the normal and expected time of 90 days for surgical healing.

CONTACTS AND LOCATIONS:
Overall Officials: Una Lee, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Overview | Drug Overdose | CDC Injury Center. Published March 19, 2020. Accessed November 5, 2020. https://www.cdc.gov/drugoverdose/data/prescribing/overview.html
- [Background] Lee DJ, Talwar R, Ding J, Chandrasekar T, Syed K, Fonshell C, Danella J, Ginzburg S, Lanchoney T, Tomaszewski J, Trabulsi E, Reese A, Smaldone M, Uzzo R, Raman JD, Guzzo TJ. Stakeholder Perspective on Opioid Stewardship After Prostatectomy: Evaluating Barriers and Facilitators From the Pennsylvania Urology Regional Collaborative. Urology. 2020 Nov;145:120-126. doi: 10.1016/j.urology.2020.05.096. Epub 2020 Jul 22. PMID 32711014
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Khorfan R, Shallcross ML, Yu B, Sanchez N, Parilla S, Coughlin JM, Johnson JK, Bilimoria KY, Stulberg JJ. Preoperative patient education and patient preparedness are associated with less postoperative use of opioids. Surgery. 2020 May;167(5):852-858. doi: 10.1016/j.surg.2020.01.002. Epub 2020 Feb 20. PMID 32087946
- [Background] Jacobs BL, Rogers D, Yabes JG, Bandari J, Ayyash OM, Maganty A, Armann KM, Worku HA, Pace NM, Shah A, Pekala KR, Yu M, Chelly JE, Macleod LC, Davies BJ. Large reduction in opioid prescribing by a multipronged behavioral intervention after major urologic surgery. Cancer. 2021 Jan 15;127(2):257-265. doi: 10.1002/cncr.33200. Epub 2020 Oct 1. PMID 33002197
- [Background] Alter TH, Ilyas AM. A Prospective Randomized Study Analyzing Preoperative Opioid Counseling in Pain Management After Carpal Tunnel Release Surgery. J Hand Surg Am. 2017 Oct;42(10):810-815. doi: 10.1016/j.jhsa.2017.07.003. Epub 2017 Sep 8. PMID 28890331
- [Background] Syed UAM, Aleem AW, Wowkanech C, Weekes D, Freedman M, Tjoumakaris F, Abboud JA, Austin LS. Neer Award 2018: the effect of preoperative education on opioid consumption in patients undergoing arthroscopic rotator cuff repair: a prospective, randomized clinical trial. J Shoulder Elbow Surg. 2018 Jun;27(6):962-967. doi: 10.1016/j.jse.2018.02.039. Epub 2018 Mar 26. PMID 29599038
- [Background] Sabesan VJ, Chatha K, Koen S, Dawoud M, Gilot G. Innovative patient education and pain management protocols to achieve opioid-free shoulder arthroplasty. JSES Int. 2020 May 4;4(2):362-365. doi: 10.1016/j.jseint.2020.01.005. eCollection 2020 Jun. PMID 32490427
- [Background] Farley KX, Anastasio AT, Kumar A, Premkumar A, Gottschalk MB, Xerogeanes J. Association Between Quantity of Opioids Prescribed After Surgery or Preoperative Opioid Use Education With Opioid Consumption. JAMA. 2019 Jun 25;321(24):2465-2467. doi: 10.1001/jama.2019.6125. PMID 31237629
- [Background] Parsa FD, Pavlosky KK, Harbison G, Yim N, Cheng J, Marison SR Jr, Parsa AA. Effect of Preoperative Patient Education on Opioid Consumption and Well-Being in Breast Augmentation. Plast Reconstr Surg. 2020 Feb;145(2):316e-323e. doi: 10.1097/PRS.0000000000006467. PMID 31985627
- [Background] Rucinski K, Cook JL. Effects of preoperative opioid education on postoperative opioid use and pain management in orthopaedics: A systematic review. J Orthop. 2020 Jan 21;20:154-159. doi: 10.1016/j.jor.2020.01.020. eCollection 2020 Jul-Aug. PMID 32025140
- [Background] Bohringer C, Astorga C, Liu H. The Benefits of Opioid Free Anesthesia and the Precautions Necessary When Employing It. Transl Perioper Pain Med. 2020;7(1):152-157. PMID 31712783